CLINICAL TRIAL: NCT04193618
Title: Conservative Surgery for Abnormally Invasive Placenta: A New Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed M Maged, MD, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 173
Record Dates: First submitted 2019-12-08; First posted 2019-12-10 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conservative surgery for placenta accretta (Experimental)
  Interventions: Procedure: Conservative surgery for placenta accretta

INTERVENTIONS:
Procedure: Conservative surgery for placenta accretta — Uterine devasculrization and transverse compressing sutures before placental delivery

SUMMARY:
Placental borders and mapping by ultrasonography and Doppler ultrasonography (placental mapping) preop. And verified intraoperatively .

bladder peritoneal dissection till the level of internal Os Uterus is incised away from the placenta

*Baby was delivered , the uterus is exteriorised and 4-5 towel clips are applied rapidly control uterine incision site bleeding .

Twenty units of diluted oxytocin and 100 to 200 cc, 37°C of heated saline were infused from here, and then the cord was clamped .

Then we proceed to systemically devascularize the uterus with the placenta in site

* internal iliac artery distal ligation:
* broad ligament and ureteric dissection:
* uterine vessels :
* posterior uterine wall compression suture :
* The utero-ovarian anastomosis branches are spared to keep blood flowing to the uterus.
* if the bladder was not fully dissected from the anterior uterine wall , now we complete the dissection,
* anterior uterine wall compression suture :
* now , we excise the invaded , irreparable anterior wall segment, with the
* then separation of the placenta manually
* if there's still mild bleeding from the uterine placental bed another full myometrial thickness anterior or posterior uterine wall transverse sutures are applied below or above the placental bed site to control bleeding until it's deemed acceptable
* in cases with separate fundal anterior incision, the high incision is repaired in layers first to give more time to compress and monitor the lower segment
* refashioning of the Lower segment , repair transversely is usually done,

DETAILED DESCRIPTION:
Placental borders and mapping were detected carefully by ultrasonography and Doppler ultrasonography (placental mapping) preop. And verified intraoperatively ..

According to the mapping, in a subset of patients we entered the abdomen by transverse suprapubic incision; in another subset we entered the abdomen by infraumbilical midline incision which was extended to a supra umbilical one in cases with anterior placentae with high upper margin .

Followed by bladder peritoneal dissection till either the level of internal Os is reached or a level with extensive adherence and/ or invasion.

Uterus is incised away from the placenta, according to the plan we described by placental mapping.

Type of uterine incisions is determined after placental mapping. Placental borders have been identified, and incisions were made far away from placenta. J-shaped, vertical and upper transverse incisions were used .

In cases of high anterior wall placentae a fundal anterior incision is made separate from the placental invaded uterine segment that will be excised later and both incisions will be repaired separately ..

* Baby was delivered , the uterus is exteriorised and 4-5 towel clips are applied rapidly control uterine incision site bleeding .

Twenty units of diluted oxytocin and 100 to 200 cc, 37°C of heated saline were infused from here, and then the cord was clamped .

Then we proceed to systemically devascularize the uterus with the placenta in site

* internal iliac artery distal ligation: posterior pelvic peritoneum is incised and bilateral internal iliac arteries are ligated distally just before the offset of the uterine artery, to avoid collateral re-feeding of the internal iliac artery in case of proximal ligation
* broad ligament and ureteric dissection: the base of each broad ligament , both its leaflets and contents are dissected upwards , towards the utero-ovarian vessels away from the uterine lower segment , both ureters are dissected until each ureteric tunnel is identified

  , emptying the base of the broad ligament bilaterally helps apply temporary manual circumferencial pressure on cervix in cases of failed conservation and excess bleeding ,
* uterine vessels : simple or figure of 8 sutures are applied to each uterine artery and vein on each side incorporating 1 cm wide of the lateral part of the lower segment , this is done just below the placenta or 1 cm above the ureteric tunnel in cases of deep placental invasion .

In cases with extensive broad ligament invasion another high uterine vessels ligation is done to reduce bleeding from the spared utero-ovarian collaterals

* posterior uterine wall compression suture : transverse mattress suture is applied at the level of the lower most bulge of the placenta, as low as the levels of the ureteric tunnels
* The utero-ovarian anastomosis branches are spared to keep blood flowing to the uterus.
* if the bladder was not fully dissected from the anterior uterine wall , now we complete the dissection, noticing the bleeding is less in amount compared to cases we undertake bladder full dissection first before devascularization
* anterior uterine wall compression suture : A transverse mattress suture is placed below the placental bulge , incorporating most of the anterior uterine wall tissues , 1 cm medial to each uterine vessel ligatures

  , at a corresponding level to the posterior uterine compression suture, while avoiding incorporating the posterior uterine wall to avoid closing the cervical canal
* now , we excise the invaded , irreparable anterior wall segment, with the First inch of the incision we notice the uterine incision bleeding , in case the bleeding is low flow & brown in colour in case of proper devascularization, if the bleeding is high flow bright red we revise our ligatures then continue the excision
* then separation of the placenta manually
* if there's still mild bleeding from the uterine placental bed another full myometrial thickness anterior or posterior uterine wall transverse sutures are applied below or above the placental bed site to control bleeding until it's deemed acceptable
* in cases with separate fundal anterior incision, the high incision is repaired in layers first to give more time to compress and monitor the lower segment
* refashioning of the Lower segment , repair transversely is usually done, in cases with a wide placental invasion disc excision of a diameter 15-20 cm, if the defect is long we close the incision longitudinally, while maintaining the cervical canal patent at all times
* we observe for vaginal bleeding for 20 - 30 minutes intraoperatively before abdominal wall closure
* closure over 2 wide bore drains
* we continue administration of oxytocin postoperatively
* we continue monitoring for vaginal bleeding for the next 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Placenta accreta spectrum, with partial or total invasion With area of invasion more than 7 cm in diameter

  * patient's informed consent about the future risks of conservative management
  * pregnancy > 20 weeks

Exclusion Criteria:

* * deeply pelvic placenta accreta spectrum cases with cervical invasion , by transvaginal ultrasound cervical length less than 21 mm

  * cases with total invasion in which the area of invasion is more than 20 min diameter
  * patient refusing conservative management and opting for hysterectomy
  * medical comorbidities making massive hemorrhage more likely such as coagulopathies
  * patient is in active antepartum hemorrhage

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-03-06 (Actual)

PRIMARY OUTCOMES:
intraoperative blood loss | during the operation
  Blood loss = estimated blood volume (EBV) x preoperative hematocrit - postoperative hematocrit/preoperative hematocrit another method by weighing the towels and dressings before and after the procedure and adding the volume of fluid inside the suction apparatus

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No